CLINICAL TRIAL: NCT00166777
Title: Effect of Hip Adduction Combination With Knee Extension Exercise on Morphology of Quadriceps Muscles, Pain and Functional Outcomes in Patients With PFPS
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Educational/Counseling/Training
Other Study IDs: 9461700808
Record Dates: First submitted 2005-09-11; First posted 2005-09-14 (Estimated); Last update posted 2006-09-11 (Estimated); Status verified 2005-08

CONDITIONS: Patellofemoral Syndrome
MeSH Terms: conditions — Patellofemoral Pain Syndrome | interventions — Exercise

INTERVENTIONS:
Procedure: exercise training

SUMMARY:
Quadriceps retraining, especially the vastus medialis oblique muscle strengthening, plays an important role in clinical management of patellofemoral pain syndrome. Vastus medialis oblique muscle roles as a dynamic stabilizer during the functional knee movement. It can generate a medial pulling force to patella against the lateral pulled by vastus lateralis. Thus it improves the patellofemoral joint compression force, reduces the knee pain, increases functional abilities, and patients' quality of life.

Could vastus medialis oblique be isolation by way of specific exercise without or minimize the recruitment of vastus lateralis？ According to human anatomy, vastus medialis oblique muscle origin from hip adductor magnus tendon, thus if incorporate hip adduction with knee extension as a selective means of training needs more researches. However, literature search shows that there are only a lot of EMG studies, so we need further clinical research to prove the treatment effect of this kind of strategy.

The purpose of the study is to investigate the treatment effects of hip adduction combine knee extension exercise in patients with patellofemoral pain syndrome. We use muscle morphology of quadriceps muscle, pain, and functional abilities as the main outcome measures. Besides, we will make further compare with traditional knee extension exercise. The first hypothesis of the study is that patients with patellofemoral pain syndrome will get improvement in muscle morphology of quadriceps muscle, pain, and functional abilities after hip adduction combine knee extension exercise training . The second hypothesis is that patients with patellofemoral pain syndrome who receive hip adduction combine knee extension exercise training will get more improvement in muscle morphology of quadriceps muscle, pain, and functional abilities than patients who receive traditional knee extension exercise training.

90 patients with patellofemoral pain syndrome who less than 50 years old will be included in this study, and randomly distributed to hip adduction combine knee extension exercise group, knee extension exercise group, and control group. Following 8 weeks exercise training by an experimental physical therapist, ultrasound measurement of muscle thickness and cross-sectional area of vastus medialis oblique muscle, vastus lateralis muscle, and rectus femoris muscle component of quadriceps, 10cm-VAS patellofemoral joint pain evaluation, including VAS-U, VAS-W, and VAS-activity, and Lysholm scale scores will be measured. A two-way mixed ANOVA will be used to compare the mean differences between theses three groups.

The study is aimed to provide an clinical evidence for evidence-based practice of rehabilitation in patients with patellofemoral pain syndrome.

ELIGIBILITY:
Inclusion Criteria:

* patients with unilateral or bilateral patellofemoral pain syndrome:

  1. age <50 y/o
  2. have anterior or retropatellar knee pain on at least 2 of the following activities: prolonged sitting, ascending or descending stairs, squatting, running, kneeling, hopping/jumping
  3. have anterior or retropatellar knee pain on at least 2 of the following evaluations: patellar palpation, resisted knee extension, patellar compression
  4. have symptoms for at least 1 month, and pain level >3cm on a VAS scale

Exclusion Criteria:

1. have severe knee pain (>8cm on a VAS scale) or referred pain
2. recent history (within 3 months) of medical therapy for pain relief
3. have history of knee surgery
4. have central or peripheral neurological pain
5. have severe knee deformity or malalignment of lower extremities
6. have regular exercise habits (15-20 mins/time, >3times/week)

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90
Dates: Start 2005-09; Study Completion 2006-06

PRIMARY OUTCOMES:
muscle morphology of quadriceps
pain serverity
functional ability

CONTACTS AND LOCATIONS:
Overall Officials: MH Jan, master, Study Chair — National Taiwan Uneversity Hospital
Locations (1):
- NTU, Taipei, Taiwan